CLINICAL TRIAL: NCT01228955
Title: Yoga Intervention for Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Debra Friedman, Division Director, Pediatric Hematology/Oncology, Vanderbilt University Medical Center
Other Study IDs: 091309
Record Dates: First submitted 2010-10-15; First posted 2010-10-27 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cancer Survivors; Yoga

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Yoga Group: Group will enter a 10 week yoga class

SUMMARY:
Impaired health related quality of life (HRQOL) including fatigue, problems with sleep and psychosocial well being (physical, emotional, and spiritual) have been noted in adult cancer survivors. Physical domain is one of the most common measured indicators of HRQOL. Despite the tremendous implications of having an impaired QOL, few studies have staged interventions aimed at improving HRQOL in a heterogeneous group of cancer survivors. There is little literature examining whether a yoga intervention is feasible in a heterogeneous group of cancer survivors.

The proposed research will utilize Vanderbilt Ingram Cancer Center (VICC), Nashville General Hospital (NGH) and REACH for Survivorship program for a pilot study. The investigators will see if a study using a broad range of diagnoses is feasible for a Yoga Intervention.

DETAILED DESCRIPTION:
The Yoga Program

The yoga intervention will be developed by a certified yoga instructor. The yoga instructors teaching the classes will undergo training before teaching classes; all classes will embody the same positions and techniques. Based on Tantric Hatha yoga techniques, the intervention will incorporate physical stretches and poses, breathing exercises and meditation. All exercises will be done in a seated or reclined position. Yoga positions will focus on breathing exercises and basic stretching and will be at the easy or basic level. Yoga positions to be utilized in the intervention are located in the Appendix. Classes will include instruction on practicing the techniques taught in the classes at home.

The yoga instructors utilized in this study are certified in yoga instruction. The classes will be held over a period of 60 minutes in a quiet, dimly lit conference room at Gilda's Club and at Nashville General Hospital. The classes will combine physical postures (asanas), breathing (pranayama) and deep relaxation (savsana). It will be made clear that participants should not practice any pose that causes or exacerbates any discomfort. Yoga poses will be modified based on participants needs. Individual poses will be held from 20 seconds to 5 minutes depending on the poses. Classes will begin slowly and progress; adding poses to the same sequence, breath techniques and restorative poses for each class over the 10 weeks. Modifications and pose variations will be used to make the class appropriate for each individual. Chairs, yoga props, and a wall will be used to assist in poses. The class will consist of the following outline:

5 Minutes: Centering, Relaxation, Body Scan

* Seated (Sukasana, Simple Cross Legged Pose)
* Reclined (Savasana, Relaxation Pose)

  10 minutes: Breathing techniques
* Diaphramic breathing (belly breath)
* Ujjayi breathing (builds heat and is an audible breath)
* Kapalabhati breathing (pumping breath)
* Nadi Sodhana breathing (alternate nostril breath)

  10 minutes: Warming spine and body
* Cat/Cow
* Twists
* 1/2 Sun Salutations and variations

  15 minutes: Strength building and stretching poses
* Hamstring Opener (reclined)
* Downward Dog (at wall or on floor)
* Lunges (at wall, with chair or with no props)
* Bridge Pose
* Locust Pose (with variations)

  5 minutes: Restorative Poses
* Supported Bridge Pose
* Supported Child's Pose
* Supported Forward Twist
* Legs up Wall
* (rotate restorative poses throughout 10 weeks)

  5 minutes:
* Savasana (final relaxation)

  5 minutes:
* Mindfulness Meditation

More details about the positions are located in the Appendix.

Study Instruments

Short Form 36 (MOS SF-36): The MOS SF-36 contains eight individual scales from which we will generate the Physical Component (PCS) and the Mental Component Summary (MCS) scores. The eight scales include physical functioning, role function-physical, bodily pain, social functioning, mental health, role function-emotional, vitality and general health perceptions [33]. The MOS SF 36 has been validated in the general population and population norms have been established for comparison between specific groups. Each scale is scored from 0-100, with 100 being the most favorable score. The SF-36 has been validated in the general population and population norms have been established for comparison between specific groups. The summary scales have been standardized to a reference normal healthy population, with a mean score of 50 and deviation of 10 points. Within the SF-36 is a 4 item Vitality scale which can be used to determine the presence or absence of fatigue.

Brief Symptom Inventory-The BSI is a short 53 item instrument designed to measure three dimensions of psychological distress - somatization, depression and anxiety. Raw scores are converted to T scores on the basis of normative data. The T scores are then dichotomized, in which a T score 63 classified a respondent as having psychological distress.

Survivor Questionnaire: A self-report questionnaire will be used to ascertain all demographic and historical information on race, age, income, education, current and past employment status, and current and past marital status. Current medical conditions will be selected by the participant from checklist including major medical conditions including secondary malignancy, cardiac, pulmonary and thyroid dysfunction. In addition, participants will be asked to list their current medications such as thyroid replacement, immunosuppressants, and anti-depressants. Lifetime smoking and alcohol habits will also be quantified, as well as reproductive history.

ELIGIBILITY:
Inclusion Criteria:

* Survivor population
* Adults (18 years of age or above)
* Patients treated for any cancers between the ages of 18 and 65 years of age
* Received and concluded cancer treatment anytime from January 1, 2000 up to 1 month before start date of study
* Received cancer treatment and care at either Vanderbilt-Ingram Cancer Center (VICC) or Nashville General Hospital (NGH) or are currently receiving cancer survivorship care at the Vanderbilt REACH for Survivorship Clinic
* Obtain *medical clearance to perform light exercise from primary care physician, oncologist or health care provider at REACH for Survivorship clinic (medical clearance needs to be obtained at least 2 weeks prior to starting yoga class).
* Have completed, if ever received, any chemotherapy treatment from January 1, 2000 up to 1 month before start date of study
* Patients with lymphedema due to cancer surgery/treatment are eligible
* Alive without evidence of recurrent disease
* Without evidence of a subsequent malignancy following initial cancer diagnosis
* Provide informed consent
* Should be able to sit on chair/floor and recline without assistance
* Can read and understand English
* Can have past experience with yoga or meditation

Exclusion Criteria:

* Enrolled or attending a yoga class at time of recruitment
* Currently receiving active treatment for cancer
* Currently not in remission
* Have any additional health concerns such as brain metastases or ventricular-peritoneal shunts at time of participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivors of Adult or Pediatric Cancer
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of Cancer Survivors interested and willing to participate in a 10 week yoga class at Vanderbilt Ingram Cancer Center (VICC) and at Nashville General Hospital | 12 months
  The investigators will be opening up an hourly yoga class for 10 weeks to all cancer survivors at VICC and at Nashville General Hospital

SECONDARY OUTCOMES:
Levels of Fatigue using the SF-36 and Psychological Distress using BSI-18 | 12 months
  Participants in the Yoga Study will be asked to complete the SF-36 and BSI-18 at three different time points in the study. Prior to start of a yoga class, at the end of the 10 week yoga class and 3 months after the completion of the yoga class.

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Friedman, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No